CLINICAL TRIAL: NCT01380496
Title: Randomized, 3-Way Crossover, Comparative Bioequivalence Study of Par Pharmaceutical Inc. (USA) and Oclassen Pharmaceuticals Inc. (USA)(Monodox(R)) Doxycycline Monohydrate Equivalent to 100 mg Doxycycline Administered as a Single Dose of 100 mg In Healthy Adult Males Under Fasting and Fed Conditions
Brief Title: Bioequivalence Study of Doxycycline Monohydrate Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: Anapharm (Industry)
Responsible Party: Alfred Elvin/Director of Biopharmaceutics, Par Pharmaceutical Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 99118
Record Dates: First submitted 2008-04-01; First posted 2011-06-27 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: To Determine Bioequivalence Under Fed Conditions
Keywords: bioequivalence; doxycycline monohydrate; fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- B (Active Comparator): Subjects received the Oclassen Pharmaceuticals Inc. formulated product.
  Interventions: Drug: doxycycline monohydrate
- C (Active Comparator): Subjects received the Oclassen Pharmaceuticals Inc. formulated product.
  Interventions: Drug: doxycycline monohydrate
- A (Experimental): Subjects received the Par formulated product
  Interventions: Drug: doxycycline monohydrate

INTERVENTIONS:
Drug: doxycycline monohydrate — tablet, 100 mg, single, oral dose
  Other Names: Monodox(R)
  Arms: A
Drug: doxycycline monohydrate — Capsule, 100 mg, single, oral dose
  Other Names: Monodox (R)
  Arms: B
Drug: doxycycline monohydrate — Capsule, 100 mg, single, oral dose
  Other Names: Monodox(R)
  Arms: C

SUMMARY:
The purpose of this study is to compare the single-dose bioequivalence of Par and Oclassen doxycycline monohydrate 100 mg.

DETAILED DESCRIPTION:
To compare the single-dose bioequivalence of Par and Oclassen (Monodox(R)), 100 mg doxycycline under fed and fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Males, non-smokers, between 18-55 years of age
* Subjects' weight will be within 15% of their ideal weight based on the Table of "Desirable Weight of Adults", Metropolitan Life Insurance Company, 1983.
* Subjects should read, sign, and date an Informed Consent Form prior to any study procedures
* Subjects must complete all screening procedures within 28 days prior to the administration of the study medication.

Exclusion Criteria:

* Clinically significant abnormalities found during medical screening
* Any clinically significant history of ongoing gastrointestinal problems or problems known to interfere with the absorption, distribution, metabolism or excretion of drugs (e.g. chronic diarrhea, inflammatory bowel diseases).
* Clinically significant illnesses within 4 weeks of the administration of study medication.
* Abnormal laboratory test judged clinically significant.
* ECG or vital signs abnormalities (clinically significant).
* History of allergic reactions to doxycycline or other related drugs (e.g., chlortetracycline, demeclocycline, minocycline and tetracycline).
* History of allergic reactions to heparin.
* Any food allergies, intolerances, restrictions, or special diet which in the opinion of the medical sub-investigator, contraindicates the subject's participation in this study.
* Positive urine drug screen (see section VIII) at screening
* Positive testing for hepatitis B, hepatitis C or HIV screening.
* Use of an investigational drug or participation in an investigational study, within 30 days prior to administration of the study medication.
* Recent donation of plasma (500 mL) within 7 days or recent donation or significant loss of whole blood (450 mL) with 56 days prior to administration of the study medication.
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than two units of alcohol per day (1 Unit = 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%)
* Recent history of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana, pot) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP), crack) within 1 year of the screening visit.
* Subjects who have taken prescription medication 14 days preceding administration of study medication or over the counter products 7 days preceding administration of study medication, except for topical products without systemic absorption.
* Subjects who have taken any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to administration of the study medication (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine).
* Subjects who have undergone clinically significant surgery 4 weeks prior to the administration of the study medication.
* Any reason which, in the opinion of the medical sub-investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 1999-11; Primary Completion 1999-11 (Actual); Study Completion 1999-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence
  Comparable food effect; The ratio of least-squares meansof the test to reference of AUCo-t, AUC -inf and Cmax should be within 80% to 125%.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Masson, Pharm D., Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Sainte-Foy, Quebec, Canada